CLINICAL TRIAL: NCT05807178
Title: Stabilization of Circadian Rhythms in Delirious ICU Patients Through Light Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Head of the Department of Anesthesiology and Intensive Care Medicine (CCM/CVK), Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIRCA-MED-WP2
Record Dates: First submitted 2023-02-23; First posted 2023-04-11 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Circadian Dysrhythmia

STUDY DESIGN:
Intervention Model Description: Evaluation of Specific Light Algorithms (Dynamic Lightening Schedule Therapy Devices) to Maintain and Restore Circadian Melatonin Rhythmicity in Critically Ill Patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LSA-1 (Experimental): Light Scheduling Algorithm-1 (LSA-1): High circadian effective irradiances
  Interventions: Device: Dynamic Light Therapy Device, LSA-1
- LSA-2 (Active Comparator): Light Scheduling Algorithm-2 (LSA-2): Irradiance levels comparable to conventional hospital lighting (control group).
  Interventions: Device: Dynamic Light Therapy Device, LSA-2

INTERVENTIONS:
Device: Dynamic Light Therapy Device, LSA-1 — Dynamic Light Therapy
  Arms: LSA-1
Device: Dynamic Light Therapy Device, LSA-2 — Light Exposition
  Arms: LSA-2

SUMMARY:
The investigators will examine the effects of dynamic light therapy on circadian rhythms in delirious intensive care unit (ICU) patients. In a randomized controlled trial (RCT), they will investigate the effects of a specific light algorithm on rhythms of serum melatonin, clock gene expression, the proteome, and metabolome, compared to standard hospital lighting, supported by the data science algorithms to improve vital-based algorithms with light interventions.

ELIGIBILITY:
Inclusion Criteria:

* Patient capable of giving consent or additionally existing legal caregiver or authorized/spouse representative in case of non-consenting patients in the intensive care unit
* Male and female patients with age ≥ 18 years
* Expected intensive care unit stay ≥ 2 days
* Positive delirium during and up to a maximum of 30 days after study inclusion (determined by CAM-ICU, at least once per shift)

Exclusion Criteria:

* Participation in other clinical studies during the study period and ten days before
* Previous ICU treatment during the current hospital stay
* Patients with psychiatric diseases
* Patients with a history of stroke and known severe residual cognitive deficits
* Patients with a history of cardiopulmonary arrest or pulseless electric activity with cardiopulmonary resuscitation followed by therapeutic hypothermia during entire hospital stay
* Amaurosis
* History of sleep-related breathing disorders
* History or suspicion of hypoxic brain damage
* History or suspicion of elevated intracranial pressure in the last 7 days before study inclusion
* Patient has a power of attorney or patient's provision, where he/she refuses participation in any clinical trial
* The informed consent of the patient or the subject's legally acceptable representative can't be obtained in time
* History of photoallergic reactions or history of visually triggered seizures
* Severe eye diseases (e.g. retinopathy, glaucoma) or high sensitivity to bright light
* Patients with liver cirrhosis
* Patients with a probability of survival <24h
* Optic neuritis within the last 3 months
* Travel across two time zones within 3 months prior to study screening
* Women who are pregnant, have a positive pregnancy test, are breastfeeding or plan to become pregnant during the course of this clinical trial
* Therapy-refractory blood coagulation disorder and inability to consent are exclusion criteria for a muscle biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-20 (Actual); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Rhythmicity of melatonin concentration | Plasma melatonin levels will be assessed for every 4 hours on day 1 and day 5 after study inclusion
  Prevalence of physiological circadian rhythmicity measured by serum melatonin concentrations.

SECONDARY OUTCOMES:
Clock genes | Clock gene expression levels will be assessed for every 4 hours on day 1 and day 5 after study inclusion.
  Prevalence of physiological circadian rhythmicity measured by expression activity of clock genes.
Metabolomics | Metabolomic measurements be assessed up to 3 (6-9) months.
  Prevalence of physiological circadian rhythmicity measured by metabolomic concentrations.
Proteomics | Proteomic measurements will be assessed up to 3 (6-9) months.
  Prevalence of physiological circadian rhythmicity measured by proteomic concentrations.
Inflammation parameters | Inflammation parameter levels will be assessed up to 3 (6-9) months.
  Prevalence of physiological circadian rhythmicity measured by inflammation parameters (cytokines, chemokines, extracellular mitochondria concentrations.
Incidence of intensive care unit delirium | Participants will be followed up until discharge from the intensive care unit (maximum up to day 5)
  Delirium will be measured with the Confusion Assessment Method for the intensive care unit (CAM-ICU), Binary scale (Positive/Negative)
Delirium-free days in the intensive care unit | Participants will be followed up until discharge from the intensive care unit (maximum up to day 5)
  Delirium-free days will be measured in day without positive delirium scoring (Confusion Assessment Method for the intensive care unit (CAM-ICU), Binary scale (Negative))
Delirium Severity | Participants will be followed up until discharge from the intensive care unit (maximum up to day 5)
  Delirium severity will be measured with the Intensive Care Delirium Screening Checklist (ICDSC). The higher the score the worse - higher score = higher delirium severity(ICDSC)
Depth of Sedation | Participants will be followed up until discharge from the intensive care unit (maximum up to day 5)
  Level of sedation will be measured with the Richmond Agitation-Sedation-Scale (RASS), -5 to +4, negative scores translates to a higher degree of sedation.
Level of analgesia 1 | Participants will be followed up until discharge from the intensive care unit (maximum up to day 5)
  Severity of pain will be measured with the Numeric Rating Scale (NRS). A higher score corresponds to a higher severity of pain.Score values from 0 to 10. A higher score means worse outcome.
Level of analgesia 2 | Participants will be followed up until discharge from the intensive care unit (maximum up to day 5)
  Severity of pain will be measured with the Visualized Numeric Rating Scale (NRS-V). A higher score corresponds to a higher severity of pain.Score values from 0 to 10. A higher score means worse outcome.
Level of analgesia 3 | Participants will be followed up until discharge from the intensive care unit (maximum up to day 5)
  Severity of pain will be measured with the Faces Pain Scale-Revised (FPS-R). A higher score corresponds to a higher severity of pain.Score values from 0 to 10. A higher score means worse outcome.
Level of analgesia 4 | Participants will be followed up until discharge from the intensive care unit (maximum up to day 5)
  Severity of pain will be measured with the Behavioral Pain Scale (BPS) . A higher score corresponds to a higher severity of pain.Score values from 3 to 12. A higher score means worse outcome.
Level of analgesia 5 | Participants will be followed up until discharge from the intensive care unit (maximum up to day 5)
  Severity of pain will be measured with the Behavioral Pain Scale for Non- Intubated (BPS-NI). A higher score corresponds to a higher severity of pain. A higher score corresponds to a higher severity of pain.Score values from 3 to 12. A higher score means worse outcome.
Total amount of opioids | Participants will be followed up until discharge from the intensive care unit (maximum up to day 5)
  Total amount of opioids administered per ICU treatment day will be measured in with morphine equivalents for each administered opioids.
Total amount of sedatives | Participants will be followed up until discharge from the intensive care unit (maximum up to day 5)
  Total amount of sedatives administered per ICU treatment day by dose summation for each sedative.
Duration of ventilation | Participants will be followed up until discharge from the intensive care unit (maximum up to day 5)
  Duration of invasive and non-invasive ventilation in hours
ICU length of stay | Participants will be followed up until ICU discharge, an expected average of 3 days.
  ICU length of stay will be measured in days
Hospital length of stay | Participants will be followed up until hospital dischargean expected average of 7 days.
  Hospital length of stay will be measured in days
Sepsis | Participants will be followed up until discharge from the intensive care unit (maximum up to day 5)
  Does patient fulfil sepsis criteria (Yes/No)
Septic shock | Participants will be followed up until discharge from the intensive care unit (maximum up to day 5)
  Does patient fulfil criteria for septic shock (Yes/No)
Sequential Organ Failure Assessment (SOFA-Score) | Participants will be followed up until discharge from the intensive care unit (maximum up to day 5)
  Predicts ICU mortality based on lab results and clinical data. . Score values between 0 and max. 24. Higher scores mean worse outcome.
Simplified Acute Physiology Score (SAPS II) | Participants will be followed up until discharge from the intensive care unit (maximum up to day 5)
  Estimates mortality in ICU patients, comparable to APACHE II.Score values between 0 and max. 163. Higher scores mean worse outcome.
Therapeutic Intervention Scoring System (TISS-28) | Participants will be followed up until discharge from the intensive care unit (maximum up to day 5)
  The Simplified Therapeutic Intervention Scoring System TISS-28 consists of 28 items. It is intended to accurately measure the level of care required for a patient in the Intensive Care Unit (ICU). Score values between 0 and max. 78. Higher scores mean higher level of required care for ICU patients.
Acute Physiological and Chronic Health Evaluation 2 Score (APACHE II) | Participants will be followed up until discharge from the intensive care unit (maximum up to day 5)
  The Acute Physiology and Chronic Health Evaluation (APACHE II) is a severity score and mortality estimation tool developed from a large sample of ICU patients in the United States.. Score values between 0 and max. 71. Higher scores mean worse outcome.
Medical Research Council (MRC) Score | Participants will be followed up until discharge from the intensive care unit (maximum up to day 5)
  The muscle scale grades muscle power on a scale of 0 to 5 (5= Muscle contracts normally against full resistance.; 0 = No movement is observed).
Hand strength measurements | Participants will be followed up until discharge from the intensive care unit (maximum up to day 5)
  Hand grip strength is measured with a dynometer.
Intensive Care Mobility Scale | Participants will be followed up until discharge from the intensive care unit (maximum up to day 5)
  To record the patient's highest level of mobility in the Intensive Care Unit. Scale from 0 to 10. 0 meaning no movement and 10 mean walking independently.
FIM Score (Functional Independence Measure) | Participants will be followed up until discharge from the intensive care unit (maximum up to day 5)
  FIM™ is comprised of 18 items, grouped into 2 subscales - motor and cognition. Each item is scored on a 7 point ordinal scale, ranging from a score of 1 to a score of 7. The higher the score, the more independent the patient is in performing the task associated with that item
Mean blood glucose (mg/dl) | Participants will be followed up until discharge from the intensive care unit (maximum up to day 5)
  Plasma glucose (PG) levels are determined by taking a blood sample from participants. It can be measured in mg/dL.
Blood glucose variability (SD in mg/dl) | Participants will be followed up until discharge from the intensive care unit (maximum up to day 5)
  Blood glucose variability (SD in mg/dl) represents how much glucose levels fluctuate over time from a given average.
Percentage of time in target glucose range (%) | Participants will be followed up until discharge from the intensive care unit (maximum up to day 5)
  Blood glucose levels outside the ranges listed in the blood sugar levels chart by age above are categorized as either high or low blood sugar.
Insulin requirement (IU/kg/h) | Participants will be followed up until discharge from the intensive care unit (maximum up to day 5)
  The amount of insuline is measured in units (IU).
Post Intensive Care Syndrome (PICS) | Up to 3 (6-9) months
  Binary scale (Positive/Negative). Diagnosis of "PICS" is defined by a new impairment or worsening of the health condition after intensive care unit stay and a clinically significant distress in at least one of the following outcome measurement instruments: Patient Health Questionnaires (PHQ-9, PHQ-8, PHQ-4), Generalized Anxiety Disorder Scales (GAD-2 and GAD-7), Impact of Event Scale Revised (IES-R), MiniCog, Animal Naming Test, Trail Making Test (TMT-A, TMT-B), Repeatable Battery for the Assessment of Neuropsychological Satus (RBANS), Timed Up-and-Go (TUG), Handgrip Strength, EQ-5D-5L, subjective assessment NRS, WHO Disability Assessment Schedule (WHODAS), Short Physical Performance Battery (SPPB).
Analysis of the sleep architecture measured by polysomnography 1 | Up to 3 (6-9) months
  Binary scale (Positive/Negative). All participants will be undergoing a polysomnography in the St. Hedwig hospital.
Analysis of the sleep architecture measured by polysomnography 2 | Participants will be followed up until discharge from the intensive care unit (maximum up to day 5)
  All participants will be undergoing a polysomnography one night in the Intensive Care Unit.
MCTQ (Munich Chronotype Questionnaire) | Up to 3 (6-9) months
  In this questionnaire, the typical sleep behaviour over the past 4 week will be reported
Actigraphy | Up to 3 (6-9) months
  Aktigraphy is measured by ActLumus in a time period of six weeks.
Sleep diary | Up to 3 (6-9) months
  Sleep parameter are documented by a sleep diary in a time period of six weeks.
Molecular data | Participants will be followed up until discharge from the intensive care unit (maximum up to day 5)
  Molecular data from muscle needle biopsies in the morning and evening on a study day
Physiotherapy | Participants will be followed up until discharge from the intensive care unit (maximum up to day 5)
  Physiotherapy is measured by a questionnaire.
Nutritional Therapy | Participants will be followed up until discharge from the intensive care unit (maximum up to day 5)
  Nutritional Therapy is measured by chart review.
Nutritional Therapy Complications | Participants will be followed up until discharge from the intensive care unit (maximum up to day 5)
  Nutritional Therapy Complications are measured by chart review.
Target protein intake | Participants will be followed up until discharge from the intensive care unit (maximum up to day 5)
  Rate in patient days on which the target protein intake was achieved
Adherence to the diet plan | Participants will be followed up until discharge from the intensive care unit (maximum up to day 5)
  Rate of days with adherence to the diet plan (yes/no)
Composition of the administered food | Participants will be followed up until discharge from the intensive care unit (maximum up to day 5)
  Composition of the administered food is measured by macro- and micronutrients according to documentation
Daily feeding breaks | Participants will be followed up until discharge from the intensive care unit (maximum up to day 5)
  Daily feeding breaks are measured in hours
Wheather data | Participants will be followed up until discharge from the intensive care unit (maximum up to day 5)
  Weather data are extracted from German Wheather Administration and Federal Environment Agency.
Cognition 1 | Up to 3 (6-9) months
  Cognition 1 is measured by MiniCog
Cognition 2 | Up to 6 months
  Cognition 2 is measured by Animal Naming Test
Cognition 3 | Up to 3 (6-9) months
  Cognition 3 is measured by Trail Making Tests A&B
Mental impairments | Up to 3 (6-9) months
  Mental impairments are measured using the PHQ-4. The PHQ-4 (Patient Health Questionnaire-4) is a brief, 4-item self-report tool screening for anxiety and depression symptoms, combining the PHQ-2 (depression) and GAD-2 (anxiety) scales, with scores from 0-12 indicating increasing symptom severity (Normal: 0-2, Mild: 3-5, Moderate: 6-8, Severe: 9-12). Each item asks how often in the last two weeks you've been bothered by something, with responses 0 (not at all) to 3 (nearly every day), and scores ≥3 on the first two items suggest depression, while ≥3 on the last two suggest anxiety, warranting further clinical assessment.
Quality of life 1 | Up to 3 (6-9) months
  Quality of life 1 is measured by EQ-5D-5L. The EQ-5D-5L is a widely used patient-reported outcome (PRO) tool measuring health-related quality of life with five dimensions (Mobility, Self-care, Usual Activities, Pain/Discomfort, Anxiety/Depression), each having five severity levels (no to extreme problems) An EQ-5D-5L result describes health status in 5 dimensions on a 5-point scale (none to extreme problems) and is summarized into a single index value (usually 0 to 1), with 1 representing perfect health, supplemented by a visual analog scale (EQ VAS) value for self-assessment of health.
Quality of life 2 | Up to 3 (6-9) months
  Quality of life 2 is measured by WHODAS 2.0. The WHODAS (World Health Organization Disability Assessment Schedule) 2.0 12-item version is a standardized, cross-cultural tool measuring health and disability by assessing difficulties in six core domains (cognition, mobility, self-care, getting along, life activities, participation) over the past 30 days, and contains 2 questions per domain. WHODAS 2.0 uses a 1-5 Likert scale (none to extreme difficulty) for its items, with scores summed and converted to a 0-100 standardized score (higher is worse), offering simple addition for general scoring or complex Item Response Theory (IRT) for weighted domain scores, with a threshold of >10 (12-item) indicating top 10% disability, all to assess disability across six domains.
Mortality | Up to 6 months
  Mortality is measured by statistical data.

OTHER OUTCOMES:
Circadian analyzes of routine high-output clinical data (Working package 1) | Before the start of this investigation
  Relevant clinical data (routine and study data), which are associated with circadian rhythmicity

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Charite University, Berlin, Germany
Locations (2):
- Germany (2):
  - Department of Anesthesiology and Intensive Care Medicine (CCM/CVK), Campus Charité Mitte, Berlin
  - Department of Anesthesiology and Intensive Care Medicine (CCM/CVK), Campus Virchow Klinikum, Berlin

IPD SHARING:
Plan to Share IPD: No